CLINICAL TRIAL: NCT05970848
Title: Washing Pipe with a Spray Nozzle for Topical Airway Anesthesia Using the Spray-as-You-Go Technique During Flexible Bronchoscopy: a Randomized Control Trial
Brief Title: Washing Pipe with a Spray Nozzle for Topical Anesthesia During Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Clinical Professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202302060RINC
Record Dates: First submitted 2023-05-24; First posted 2023-08-01 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease
Keywords: flexible bronchoscopy; topical airway anesthesia
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: Group S patients will receive topical lidocaine anesthesia via the spray nozzle by the spray as-you-go technique during flexible bronchoscopy. Group C patients will receive topical lidocaine anesthesia with the conventional method by the spray as-you-go technique during flexible bronchoscopy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomly allocated into one of the two groups by the randomization module in REDCap. Patients and outcomes assessor will be blinded to their grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group S (Experimental): Group S patients will receive topical lidocaine anesthesia via the spray nozzle by the spray as-you-go technique during flexible bronchoscopy.
  Interventions: Device: Washing Pipe With a Spray Nozzle
- Group C (No Intervention): Group C patients will receive topical lidocaine anesthesia with the conventional method by the spray as-you-go technique during flexible bronchoscopy.

INTERVENTIONS:
Device: Washing Pipe With a Spray Nozzle — Administration of topical airway anesthesia via a washing pipe with a spray nozzle using the spray-as-you-go technique
  Arms: Group S

SUMMARY:
The goal of this randomized control trial is to evaluate the effectiveness and safety of using a spray nozzle, compared to the conventional method, for topical anesthesia by the spray-as-you-go technique in reducing cough frequency, improving cough, discomfort, tolerance, satisfaction, reducing the dosage of lidocaine consumption of patients during flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. A planned flexible bronchoscopy
3. Being able to communicate with Mandarin Chinese or Taiwanese Hokkien

Exclusion Criteria:

1. are unwilling to join the study
2. have tracheostomy or are intubated
3. will receive intravenous anesthesia during flexible bronchoscopy
4. known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Cough rate | Through the duration of the bronchoscopy exam, an average of 30 min
  The bronchoscopy procedure will be audio-taped throughout and cough counting will be recorded by an investigator blinded to the patient information and grouping. The cough rate will be calculated as total cough counts divided by procedure time in minute.

SECONDARY OUTCOMES:
Procedure time | Through the duration of the bronchoscopy exam, an average of 30 min
  The duration (minute) of the bronchoscopic procedure
Lidocaine dosage | Through the duration of the bronchoscopy exam, an average of 30 min
  Total lidocaine doses dispensed during the bronchoscopic procedure
Patient tolerance | Through the duration of the bronchoscopy exam, an average of 30 min
  Using a visual analogue scale from 0 to 10 to indicate patient tolerance of the bronchoscopy
Patient satisfaction | Through the duration of the bronchoscopy exam, an average of 30 min
  Using a visual analogue scale from 0 to 10 to indicate patient satisfaction of the bronchoscopy
Adverse events | Through the duration of the bronchoscopy exam, an average of 30 min
  Development of adverse events during the bronchoscopic procedure, such as bleeding and oxygen desaturation

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Criner GJ, Eberhardt R, Fernandez-Bussy S, Gompelmann D, Maldonado F, Patel N, Shah PL, Slebos DJ, Valipour A, Wahidi MM, Weir M, Herth FJ. Interventional Bronchoscopy. Am J Respir Crit Care Med. 2020 Jul 1;202(1):29-50. doi: 10.1164/rccm.201907-1292SO. PMID 32023078
- [Background] Mohan A, Madan K, Hadda V, Tiwari P, Mittal S, Guleria R, Khilnani GC, Luhadia SK, Solanki RN, Gupta KB, Swarnakar R, Gaur SN, Singhal P, Ayub II, Bansal S, Bista PR, Biswal SK, Dhungana A, Doddamani S, Dubey D, Garg A, Hussain T, Iyer H, Kavitha V, Kalai U, Kumar R, Mehta S, Nongpiur VN, Loganathan N, Sryma PB, Pangeni RP, Shrestha P, Singh J, Suri T, Agarwal S, Agarwal R, Aggarwal AN, Agrawal G, Arora SS, Thangakunam B, Behera D; Jayachandra; Chaudhry D, Chawla R, Chawla R, Chhajed P, Christopher DJ, Daga MK, Das RK, D'Souza G, Dhar R, Dhooria S, Ghoshal AG, Goel M, Gopal B, Goyal R, Gupta N, Jain NK, Jain N, Jindal A, Jindal SK, Kant S, Katiyar S, Katiyar SK, Koul PA, Kumar J, Kumar R, Lall A, Mehta R, Nath A, Pattabhiraman VR, Patel D, Prasad R, Samaria JK, Sehgal IS, Shah S, Sindhwani G, Singh S, Singh V, Singla R, Suri JC, Talwar D, Jayalakshmi TK, Rajagopal TP. Guidelines for diagnostic flexible bronchoscopy in adults: Joint Indian Chest Society/National College of chest physicians (I)/Indian association for bronchology recommendations. Lung India. 2019 Jul;36(Supplement):S37-S89. doi: 10.4103/lungindia.lungindia_108_19. PMID 32445309
- [Background] Madan K, Mohan A, Agarwal R, Hadda V, Khilnani GC, Guleria R. A survey of flexible bronchoscopy practices in India: The Indian bronchoscopy survey (2017). Lung India. 2018 Mar-Apr;35(2):98-107. doi: 10.4103/lungindia.lungindia_417_17. PMID 29487243
- [Background] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Background] Kim SY, Lee HJ, Lee JK, Park TY, Heo EY, Kim DK, Chung HS, Lee HW. Association between oxygen saturation level during bronchoscopy and post-bronchoscopy adverse events: a retrospective cohort study. Respir Res. 2022 Jun 2;23(1):144. doi: 10.1186/s12931-022-02063-0. PMID 35655299
- [Background] Fujimoto K, Ishiwata T, Kasai H, Terada J, Shionoya Y, Ikari J, Kawata N, Tada Y, Tsushima K, Tatsumi K. Identification of factors during bronchoscopy that affect patient reluctance to undergo repeat examination: Questionnaire analysis after initial bronchoscopy. PLoS One. 2018 Dec 6;13(12):e0208495. doi: 10.1371/journal.pone.0208495. eCollection 2018. PMID 30521615
- [Background] Ling IT, Piccolo F, Mulrennan SA, Phillips MJ. Posture influences patient cough rate, sedative requirement and comfort during bronchoscopy: An observational cohort study. Cough. 2011 Nov 10;7:9. doi: 10.1186/1745-9974-7-9. PMID 22074355
- [Background] Antoniades N, Worsnop C. Topical lidocaine through the bronchoscope reduces cough rate during bronchoscopy. Respirology. 2009 Aug;14(6):873-6. doi: 10.1111/j.1440-1843.2009.01587.x. PMID 19703068
- [Background] Cai Y, Chen L, Dong D, Ye M, Jin X, Liu F. The utility of a multi-orifice epidural catheter when using the "Spray-as-You-Go" technique for topical Airway Anesthesia during Flexible Bronchoscopy, a randomised trial. J Clin Monit Comput. 2023 Feb;37(1):55-62. doi: 10.1007/s10877-022-00856-8. Epub 2022 Apr 20. PMID 35441943
- [Background] Venkatnarayan K, Devaraj U, Krishnaswamy UM, Ramachandran P, Thomas T, D'Souza G. Comparison of spray catheter with "spray-as-you-go" technique for airway anesthesia during flexible bronchoscopy - A randomized trial. Lung India. 2020 Sep-Oct;37(5):384-388. doi: 10.4103/lungindia.lungindia_528_19. PMID 32883896
- [Background] Yildirim F, Ozkaya S, Yurdakul AS. Factors affecting patients' comfort during fiberoptic bronchoscopy and endobronchial ultrasound. J Pain Res. 2017 Mar 29;10:775-781. doi: 10.2147/JPR.S118047. eCollection 2017. PMID 28435314
- [Background] Kobayashi F, Saraya T, Oda M, Sakuma S, Watanabe M, Takata S, Tamura M, Takakura H, Nakamoto K, Honda K, Ohkuma K, Mikura S, Inoue M, Hirata A, Kurokawa N, Shirai T, Aso K, Noda A, Miyaoka C, Yoshida Y, Ishikawa N, Morita K, Ieki E, Nakajima H, Ishii H, Takizawa H. Novel predictive factors for patient discomfort and severe cough during bronchoscopy: A prospective questionnaire analysis. PLoS One. 2020 Oct 19;15(10):e0240485. doi: 10.1371/journal.pone.0240485. eCollection 2020. PMID 33075060
- [Background] Lechtzin N, Rubin HR, White P Jr, Jenckes M, Diette GB. Patient satisfaction with bronchoscopy. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1326-31. doi: 10.1164/rccm.200203-231OC. Epub 2002 Jul 19. PMID 12406852